CLINICAL TRIAL: NCT05150769
Title: Preferences of Vaccination for COVID-19 Among University Students and Staff: A Discrete Choice Experiment
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Esther Wai Yin Chan, Associate Professor, The University of Hong Kong
Other Study IDs: DCE_COVID-19
Record Dates: First submitted 2021-12-08; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Preference, Patient
MeSH Terms: conditions — Patient Preference

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
From March 2021, COVID-19 vaccines have been made available to Hong Kong residents, first to priority groups including healthcare professionals and the elderly, and later to all adults and adolescents. Vaccinated individuals are generally exempted from mandatory regular out-of-pocket antigen testing. Vaccinated individuals of university halls and colleges of The University of Hong Kong (HKU) will also be exempted from mandatory weekly antigen testing. Freedom of choice is highly respected in the HKU community and as such, we would like to better understand the decision-making process among members of the HKU community. The anonymised results of this independent research study will help us understand preferences among the HKU community and inform on future vaccination planning policies.

Objectives: To elicit HKU staff and students' preferences and their willingness-to-pay (WTP) for COVID-19 vaccination in Hong Kong

Design: An online cross-sectional internet-based questionnaire with a discrete choice experiment (DCE) design distributed via email. All current students and staff from the University of Hong Kong are eligible to participate in the study

Main outcome measures: Preferences for the efficacy of protecting against infection, against severe disease manifestations, duration of protection, risk of adverse events, incentives, and out-of-pocket costs

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Fluent in English
* Students and staff of The University of Hong Kong

Exclusion Criteria:

* Individuals who are younger than 18 years old
* Individuals who are unwilling to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: University students and staff working at university
Sampling Method: Non-Probability Sample
Enrollment: 3423 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2021-09-21 (Actual)

PRIMARY OUTCOMES:
Preferences for efficacy of protection against infection | At baseline
Preferences for efficacy of protection against severe disease manifestations | At baseline
Preferences for duration of protection | At baseline
Preferences for risk of adverse events | At baseline
Preferences for incentives | At baseline
Preferences for out-of-pocket cost | At baseline

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong